CLINICAL TRIAL: NCT05139758
Title: Correlation Between Anthropometric Measurements And Balance IN Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim Ali Ibrahim, Ahmed Ibrahim Ali Ibrahim Mohamed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: P.T.REC/012/003333
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Anthropometric Measurements&Balance IN CP Children
Keywords: ANTHROPOMETRIC MEASUREMENTS; BALANCE; CEREBRAL PALSY
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hemiplegic cp (Experimental): it will be classified into two subgroups according to body mass index to underweight and healthy weight .
  Interventions: Diagnostic Test: Biodex Balane System
- diplegic cp (Experimental): it will be classified into two subgroups according to body mass index to underweight and healthy weight .
  Interventions: Diagnostic Test: Biodex Balane System

INTERVENTIONS:
Diagnostic Test: Biodex Balane System — The Biodex balance system will be used for the assessment of static and dynamic balance of all children in the current study.

SUMMARY:
The purpose of the current study is to evaluate the correlation between anthropometric measurement (weight, height and BMI) and balance in children with cerebral palsy.

DETAILED DESCRIPTION:
* The European Society for Clinical Nutrition and Metabolism has pointed out that under-nutrition can led to change in body composition (e.g. depletion of body fat mass) and diminished function and outcome.
* The prevalence of under-nutrition in children with CP varies from 3.9 per cent to 71 percent mainly depending on the method of assessment, the severity of motor involvement and feeding problems.
* Studies indicate that children and adults with both mild and severe forms of CP have postural impairments. Dysfunctional posture control interferes with the activities of daily life .
* Children with CP may have impaired muscle tone and abnormal postural control, both of which affect functional balance capacity.
* There were associations between excess body weight and values below normal in some balance conditions, indicating that the anthropometric indicators interfered in the children's postural balance.

There were associations between excess body weight and values below normal in some balance conditions, indicating that the anthropometric indicators interfered in the children's postural balance.

Knowledge of anthropometric measurements and whether they affect balance in children with CP will help clinicians to develop treatment programs which in turn will improve the overall balance and functional abilities of children with CP.

* Childeren age will be ranged from 8-12 years and on level Ⅰ and Ⅱ on Growth Motor Function Classification System
* Weight would be obtained on a digital scale (UNISCALE )
* Standing height was measured using a stadiometer with a fixed vertical backboard and an adjustable head piece.
* CDC 2000 charts will be used to measure BMI
* The Biodex balance system will be used for the assessment of static and dynamic balance of all children

ELIGIBILITY:
Inclusion Criteria:

1. Their age will be ranged from 8 to 12 years.
2. The degree of their spasticity will be ranged from 1 to 2 according to Modified Ashworth' Scale.
3. They will be on level Ⅰ and Ⅱ on Growth Motor Function Classification System (GMFCS).
4. They will be able to stand without the use of an assistive device
5. Children can follow instructions and understand given orders.

Exclusion Criteria:

1. Severe visual or hearing impairment.
2. Fixed deformities or surgical interventions in the lower extremities.
3. Botulinum toxin injections in the last 6 months.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Is there a correlation between anthropometric measurements and balance in children with cerebral palsy? | 6 months
  The purpose of the current study is to evaluate the correlation between anthropometric measurement (weight, height and BMI) and balance in children with cerebral palsy.

CONTACTS AND LOCATIONS:
Overall Officials: Gehan El meniawy, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication
Access Criteria: IPD will be shared with researchers

REFERENCES:
- [Background] Adamu AS, Sabo UA, Gwarzo GD, Belonwu RO. Nutritional status in cerebral palsy: A Cross-sectional comparative survey of children in Kano, Nigeria. Niger Postgrad Med J. 2018 Jul-Sep;25(3):156-160. doi: 10.4103/npmj.npmj_67_18. PMID 30264766
- [Background] Alvarez Zaragoza C, Vasquez Garibay EM, Garcia Contreras AA, Larrosa Haro A, Romero Velarde E, Rea Rosas A, Cabrales de Anda JL, Vega Olea I. Bone mineral density and nutritional status in children with quadriplegic cerebral palsy. Arch Osteoporos. 2018 Mar 4;13(1):17. doi: 10.1007/s11657-018-0434-8. PMID 29504042
- [Background] Arifin N, Abu Osman NA, Wan Abas WA. Intrarater test-retest reliability of static and dynamic stability indexes measurement using the Biodex Stability System during unilateral stance. J Appl Biomech. 2014 Apr;30(2):300-4. doi: 10.1123/jab.2013-0130. Epub 2013 Jul 20. PMID 23878204
- [Background] Aydog E, Bal A, Aydog ST, Cakci A. Evaluation of dynamic postural balance using the Biodex Stability System in rheumatoid arthritis patients. Clin Rheumatol. 2006 Jul;25(4):462-7. doi: 10.1007/s10067-005-0074-4. Epub 2005 Oct 25. PMID 16247584
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Brooks J, Day S, Shavelle R, Strauss D. Low weight, morbidity, and mortality in children with cerebral palsy: new clinical growth charts. Pediatrics. 2011 Aug;128(2):e299-307. doi: 10.1542/peds.2010-2801. Epub 2011 Jul 18. PMID 21768315
- [Background] Bullock-Saxton JE. Local sensation changes and altered hip muscle function following severe ankle sprain. Phys Ther. 1994 Jan;74(1):17-28; discussion 28-31. doi: 10.1093/ptj/74.1.17. PMID 8265724
- [Background] Cumberworth VL, Patel NN, Rogers W, Kenyon GS. The maturation of balance in children. J Laryngol Otol. 2007 May;121(5):449-54. doi: 10.1017/S0022215106004051. Epub 2006 Nov 14. PMID 17105679
- [Background] Dawson N, Dzurino D, Karleskint M, Tucker J. Examining the reliability, correlation, and validity of commonly used assessment tools to measure balance. Health Sci Rep. 2018 Oct 27;1(12):e98. doi: 10.1002/hsr2.98. eCollection 2018 Dec. PMID 30623052
- [Background] Duran I, Martakis K, Rehberg M, Semler O, Schoenau E. Anthropometric measurements to identify undernutrition in children with cerebral palsy. Dev Med Child Neurol. 2019 Oct;61(10):1168-1174. doi: 10.1111/dmcn.14225. Epub 2019 Mar 29. PMID 30927269
- [Background] Gan SM, Tung LC, Tang YH, Wang CH. Psychometric properties of functional balance assessment in children with cerebral palsy. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):745-53. doi: 10.1177/1545968308316474. Epub 2008 Jul 21. PMID 18645187
- [Background] Garcia Iniguez JA, Vasquez-Garibay EM, Garcia Contreras A, Romero-Velarde E, Troyo Sanroman R. Assessment of anthropometric indicators in children with cerebral palsy according to the type of motor dysfunction and reference standard. Nutr Hosp. 2017 Mar 30;34(2):315-322. doi: 10.20960/nh.353. PMID 28421784
- [Background] Gulati S, Sondhi V. Cerebral Palsy: An Overview. Indian J Pediatr. 2018 Nov;85(11):1006-1016. doi: 10.1007/s12098-017-2475-1. Epub 2017 Nov 20. PMID 29152685
- [Background] Haapala H, Peterson MD, Daunter A, Hurvitz EA. Agreement Between Actual Height and Estimated Height Using Segmental Limb Lengths for Individuals with Cerebral Palsy. Am J Phys Med Rehabil. 2015 Jul;94(7):539-46. doi: 10.1097/PHM.0000000000000205. PMID 25299521
- [Background] Horak FB, Wrisley DM, Frank J. The Balance Evaluation Systems Test (BESTest) to differentiate balance deficits. Phys Ther. 2009 May;89(5):484-98. doi: 10.2522/ptj.20080071. Epub 2009 Mar 27. PMID 19329772
- [Background] Hurvitz EA, Green LB, Hornyak JE, Khurana SR, Koch LG. Body mass index measures in children with cerebral palsy related to gross motor function classification: a clinic-based study. Am J Phys Med Rehabil. 2008 May;87(5):395-403. doi: 10.1097/PHM.0b013e3181617736. PMID 18174849
- [Background] Jelsma J, Pronk M, Ferguson G, Jelsma-Smit D. The effect of the Nintendo Wii Fit on balance control and gross motor function of children with spastic hemiplegic cerebral palsy. Dev Neurorehabil. 2013;16(1):27-37. doi: 10.3109/17518423.2012.711781. Epub 2012 Oct 3. PMID 23030836
- [Background] Kuperminc MN, Gottrand F, Samson-Fang L, Arvedson J, Bell K, Craig GM, Sullivan PB. Nutritional management of children with cerebral palsy: a practical guide. Eur J Clin Nutr. 2013 Dec;67 Suppl 2:S21-3. doi: 10.1038/ejcn.2013.227. No abstract available. PMID 24301005
- [Background] Kurz MJ, Arpin DJ, Corr B. Differences in the dynamic gait stability of children with cerebral palsy and typically developing children. Gait Posture. 2012 Jul;36(3):600-4. doi: 10.1016/j.gaitpost.2012.05.029. Epub 2012 Jun 27. PMID 22743027
- [Background] Lara S, Graup S, Balk RS, Teixeira LP, Farias AD, Alves GB, Leiria VB. ASSOCIATION BETWEEN POSTURAL BALANCE AND ANTHROPOMETRIC INDEXES IN ELEMENTARY SCHOOLCHILDREN. Rev Paul Pediatr. 2017 Nov 13;36(1):7. doi: 10.1590/1984-0462/;2018;36;1;00011. Print 2018 Jan-Mar. PMID 29160409
- [Background] Meseguer-Henarejos AB, Sanchez-Meca J, Lopez-Pina JA, Carles-Hernandez R. Inter- and intra-rater reliability of the Modified Ashworth Scale: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2018 Aug;54(4):576-590. doi: 10.23736/S1973-9087.17.04796-7. Epub 2017 Sep 13. PMID 28901119
- [Background] McIlvain G, Tracy JB, Chaze CA, Petersen DA, Villermaux GM, Wright HG, Miller F, Crenshaw JR, Johnson CL. Brain Stiffness Relates to Dynamic Balance Reactions in Children With Cerebral Palsy. J Child Neurol. 2020 Jun;35(7):463-471. doi: 10.1177/0883073820909274. Epub 2020 Mar 23. PMID 32202191
- [Background] Minocha P, Sitaraman S, Choudhary A, Yadav R. Subjective Global Nutritional Assessment: A Reliable Screening Tool for Nutritional Assessment in Cerebral Palsy Children. Indian J Pediatr. 2018 Jan;85(1):15-19. doi: 10.1007/s12098-017-2501-3. Epub 2017 Oct 12. PMID 29022211
- [Background] Mutlu A, Livanelioglu A, Gunel MK. Reliability of Ashworth and Modified Ashworth scales in children with spastic cerebral palsy. BMC Musculoskelet Disord. 2008 Apr 10;9:44. doi: 10.1186/1471-2474-9-44. PMID 18402701
- [Background] Ogden CL, Flegal KM. Changes in terminology for childhood overweight and obesity. Natl Health Stat Report. 2010 Jun 25;(25):1-5. PMID 20939253
- [Background] Opheim A, Jahnsen R, Olsson E, Stanghelle JK. Balance in relation to walking deterioration in adults with spastic bilateral cerebral palsy. Phys Ther. 2012 Feb;92(2):279-88. doi: 10.2522/ptj.20100432. Epub 2011 Oct 27. PMID 22033070
- [Background] Oskoui M, Coutinho F, Dykeman J, Jette N, Pringsheim T. An update on the prevalence of cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2013 Jun;55(6):509-19. doi: 10.1111/dmcn.12080. Epub 2013 Jan 24. PMID 23346889
- [Background] Pascoe J, Thomason P, Graham HK, Reddihough D, Sabin MA. Body mass index in ambulatory children with cerebral palsy: A cohort study. J Paediatr Child Health. 2016 Apr;52(4):417-21. doi: 10.1111/jpc.13097. PMID 27145505
- [Background] Paulson A, Vargus-Adams J. Overview of Four Functional Classification Systems Commonly Used in Cerebral Palsy. Children (Basel). 2017 Apr 24;4(4):30. doi: 10.3390/children4040030. PMID 28441773
- [Background] Piscitelli D, Ferrarello F, Ugolini A, Verola S, Pellicciari L. Measurement properties of the Gross Motor Function Classification System, Gross Motor Function Classification System-Expanded & Revised, Manual Ability Classification System, and Communication Function Classification System in cerebral palsy: a systematic review with meta-analysis. Dev Med Child Neurol. 2021 Nov;63(11):1251-1261. doi: 10.1111/dmcn.14910. Epub 2021 May 24. PMID 34028793
- [Background] Richards CL, Malouin F. Cerebral palsy: definition, assessment and rehabilitation. Handb Clin Neurol. 2013;111:183-95. doi: 10.1016/B978-0-444-52891-9.00018-X. PMID 23622163
- [Background] Rieken R, Calis EA, Tibboel D, Evenhuis HM, Penning C. Validation of skinfold measurements and bioelectrical impedance analysis in children with severe cerebral palsy: a review. Clin Nutr. 2010 Apr;29(2):217-21. doi: 10.1016/j.clnu.2009.07.009. Epub 2009 Aug 14. PMID 19683370
- [Background] Rosenbaum PL, Palisano RJ, Bartlett DJ, Galuppi BE, Russell DJ. Development of the Gross Motor Function Classification System for cerebral palsy. Dev Med Child Neurol. 2008 Apr;50(4):249-53. doi: 10.1111/j.1469-8749.2008.02045.x. Epub 2008 Mar 1. PMID 18318732
- [Background] Simsek TT, Tuc G. Examination of the relation between body mass index, functional level and health-related quality of life in children with cerebral palsy. Turk Pediatri Ars. 2014 Jun 1;49(2):130-7. doi: 10.5152/tpa.2014.1238. eCollection 2014 Jun. PMID 26078648
- [Background] Soeters P, Bozzetti F, Cynober L, Forbes A, Shenkin A, Sobotka L. Defining malnutrition: A plea to rethink. Clin Nutr. 2017 Jun;36(3):896-901. doi: 10.1016/j.clnu.2016.09.032. Epub 2016 Oct 8. PMID 27769782
- [Background] Spittle AJ, Orton J. Cerebral palsy and developmental coordination disorder in children born preterm. Semin Fetal Neonatal Med. 2014 Apr;19(2):84-9. doi: 10.1016/j.siny.2013.11.005. Epub 2013 Dec 2. PMID 24290908
- [Background] Stevenson RD, Conaway M, Chumlea WC, Rosenbaum P, Fung EB, Henderson RC, Worley G, Liptak G, O'Donnell M, Samson-Fang L, Stallings VA; North American Growth in Cerebral Palsy Study. Growth and health in children with moderate-to-severe cerebral palsy. Pediatrics. 2006 Sep;118(3):1010-8. doi: 10.1542/peds.2006-0298. PMID 16950992
- [Background] te Velde A, Morgan C, Novak I, Tantsis E, Badawi N. Early Diagnosis and Classification of Cerebral Palsy: An Historical Perspective and Barriers to an Early Diagnosis. J Clin Med. 2019 Oct 3;8(10):1599. doi: 10.3390/jcm8101599. PMID 31623303
- [Background] Wood E, Rosenbaum P. The gross motor function classification system for cerebral palsy: a study of reliability and stability over time. Dev Med Child Neurol. 2000 May;42(5):292-6. doi: 10.1017/s0012162200000529. PMID 10855648